CLINICAL TRIAL: NCT01297738
Title: The Effect of Dietary Patterns and Diet Composition on Insulin Sensitivity and Cerebral Dopamine- and Serotonin Transporters
Brief Title: Diet, Insulin Sensitivity And the Brain
Acronym: DISAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Principal Investigator, K.E.M. Koopman, ms, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DISAB
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Obesity; Diabetes Mellitus Type 2
Keywords: diet manipulation; serotonin; dopamine; insulin sensitivity
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Meal size increase with HFHS (Experimental): On top of a healthy, eucaloric diet, study subjects consume a 40% calory surplus by consuming a liquid meal which is high in fat and sugar (Nutridrink®)
  Interventions: Other: Meal size increase with HFHS
- Meal size increase with HS (Experimental): On top of a healthy, eucaloric diet, study subjects consume a 40% calory surplus by consuming commercially available sugar-sweetened beverages. Subjects consume this caloric surplus with their meals, which results in an increase in meal size.
  Interventions: Other: Meal size increase with HS
- Meal frequency increase with HFHS (Experimental): On top of a healthy, eucaloric diet, study subjects consume a 40% calory surplus by consuming a liquid meal which has a high fat and sugar content(Nutridrink®). Subjects consume the Nutridrink 3 times a day in between meals. which results in an increase in meal frequency.
  Interventions: Other: Meal frequency increase with HFHS
- Meal frequency increase with HS (Experimental): On top of a healthy, eucaloric diet, study subjects consume a 40% calory surplus by consuming commercially available sugar-sweetened beverages. Subjects consume these sugar-sweetened beverages 3 times a day in between meals, which results in an increase in meal frequency.
  Interventions: Other: Meal frequency increase with HS
- Control group (No Intervention): Subjects will not follow any diet but their own ad-libitum, healty diet.

INTERVENTIONS:
Other: Meal size increase with HFHS — On top of a healthy, eucaloric diet, study subjects consume a 40% calory surplus by consuming a high-fat, high-sugar liquid medical food supplement (Nutridrink®). Subjects consume the Nutridrink® with their meals, which results in an increase in meal size.
  Other Names: Nutridrink
  Arms: Meal size increase with HFHS
Other: Meal size increase with HS — On top of a healthy, eucaloric diet, study subjects consume a 40% calory surplus by consuming commercially available sugar-sweetened beverages. Subjects consume these sugar-sweetened beverages with their meals, which results in an increase in meal size.
  Arms: Meal size increase with HS
Other: Meal frequency increase with HFHS — On top of a healthy, eucaloric diet, study subjects consume a 40% calory surplus by consuming a high-fat, high-sugar liquid medical food supplement (Nutridrink®). Subjects consume the Nutridrink® 3 times a day in between meals, which results in an increase in meal frequency.
  Other Names: Nutridrink
  Arms: Meal frequency increase with HFHS
Other: Meal frequency increase with HS — On top of a healthy, eucaloric diet, study subjects consume a 40% calory surplus by consuming commercially available sugar-sweetened beverages. Subjects consume these sugar-sweetened beverages 3 times a day in between meals, which results in an increase in meal frequency.
  Arms: Meal frequency increase with HS

SUMMARY:
Obesity and insulin resistance may be in part explained by an altered reward system with changes in the serotonin/dopamine system. These changes might be caused by changes in dietary habits, especially by an increased intake of liquid sugar and an increase in meal frequency. The investigators hypothesize that increasing meal frequency compared to increasing meal size and when consuming a hypercaloric high-sugar diet (HS) compared to a hypercaloric high-fat-high-sugar diet (HFHS) will result in a reduction in cerebral serotonin and dopamine transporters and in a more prominent increase in insulin resistance. In addition, the investigators hypothesize that the changes in insulin sensitivity will be independent of changes in abdominal (visceral) and liver fat and that changes in insulin sensitivity due to the dietary manipulation will co-occur with changes in insulin signaling pathways in peripheral fat and muscle tissue.

DETAILED DESCRIPTION:
Lean, healthy, young men will follow a hypercaloric HF- or HFHS diet for 6 weeks. Before and after the dietary intervention, the investigators will perform a SPECT-scan for serotonin and dopamine transporters with the radioligand [123I]FP-CIT, administered intravenously. The investigators will also perform a structural MRI for localization. Furthermore the investigators will perform a liver MRS and abdominal MRI for liver fat- and abdominal visceral fat measurement. The investigators will also perform a euglycemic, hyperinsulinemic clamp to measure insulin sensitivity and muscle- and fat biopsies to examine changes in insulin signaling pathways and fat metabolism. After the hypercaloric diet subjects will follow a hypocaloric diet until their weight is back to baseline.

ELIGIBILITY:
Inclusion Criteria:

* BMI 19-26 kg/m2
* Age 18-40 years old
* Male gender
* Caucasian
* Stable weight 3 months prior to start study participation

Exclusion Criteria:

* Abnormal oral glucose tolerance test (OGTT)
* Lipid disorders, renal disorders, thyroid disorders, elevated liver enzymes
* Use of medication
* Use of alcohol > 3/day
* Use of ecstasy, amphetamines or cocaine
* Smoking
* History of eating disorder or psychiatric disorder
* Any medical condition, intensive sports ( >3 times/week), shift work

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2011-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Cerebral binding of [123I]FP-CIT to serotonin- and dopamine transporters and correlation with changes in in vivo and ex vivo insulin sensitivity | At baseline and after 6 weeks of hypercaloric HFHS or HS diet
  Difference in cerebral binding of the radioligand [123I]FP-CIT to serotonin- and dopamine transporters before and after dietary manipulations and correlation of cerebral dopamine and serotonin transporter binding with changes in in vivo and ex vivo insulin sensitivity.

SECONDARY OUTCOMES:
Abdominal fat mass | At baseline and after 6 weeks of HFHS or HS hypercaloric diet
  Changes in accumulated amount of abdominal (visceral) and liver fat
Glucoregularoty hormones | At baseline and after 6 weeks of hypercaloric HFHS- or HS diet
  Changes in glucoregulatory hormones such as glucagon and leptin
Insulin signalling pathways | At baseline and after 6 weeks of hypercaloric HFHS- or HS diet
  Changes in insulin signalling pathways in peripheral fat and muscle tissue

CONTACTS AND LOCATIONS:
Overall Officials: Mireille JM Serlie, Dr, Study Director — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Karin EM Koopman, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Koopman KE, Caan MW, Nederveen AJ, Pels A, Ackermans MT, Fliers E, la Fleur SE, Serlie MJ. Hypercaloric diets with increased meal frequency, but not meal size, increase intrahepatic triglycerides: a randomized controlled trial. Hepatology. 2014 Aug;60(2):545-53. doi: 10.1002/hep.27149. Epub 2014 May 13. PMID 24668862